CLINICAL TRIAL: NCT03010397
Title: PROGRESS - Progression of Diabetic Retinopathy. Identification of Signs and Surrogate Outcomes
Brief Title: Progression of Diabetic Retinopathy. Identification of Signs and Surrogate Outcomes
Acronym: PROGRESS
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: IPM-2016
Record Dates: First submitted 2016-09-19; First posted 2017-01-05 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Progression of Diabetic Retinopathy. Identification of Signs and Surrogate outcomes (PROGRESS)

DETAILED DESCRIPTION:
The global aim of this study is to improve the current knowledge of diabetic retinopathy (DR) progression. We aim to characterize both functionally and morphologically initial DR stages and to identify patients at risk of progression to centre involving macular oedema (CME) and/or proliferative diabetic retinopathy (PDR). We want to identify imaging patterns and characteristics that might be used as prognostic biomarkers for DR progression.

For this, ischemia and blood-retinal barrier alteration will be assessed using non-invasive retinal imaging methodologies. SD-OCT with layer-by-layer segmentation will be performed. Furthermore, a state-of-the-art methodology with OCT-Angiography will be used for identification of areas of capillary drop-out and leakage areas will be identified on SD-OCT without the need of a dye injection. In a subgroup of patients we will study neurodegeneration patterns using multifocal ERG examination.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus according to 1985 WHO criteria
* Aged between 35 years and 80 at baseline in the retrospective period
* NPDR level < 20 (MA absent) or Mild NPDR (levels 20 to 35, based on ETDRS criteria- 7 fields CFP) at baseline
* BCVA ≥ 75 letters (≥ 20/32) at baseline (ETDRS charts)
* Informed Consent

Exclusion Criteria:

* Inadequate ocular media and/ or pupil dilatation that interfere with fundus examinations
* HbA1C > 10 % at the Screening or previous 6 months in the previous prospective study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients followed under the normal clinical practice at AIBILI Clinical Trial Centre.
  - Type 2 diabetes mellitus according to 1985 WHO criteria
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Phenotypic classification of DR in a 5-year period | 5 years
  Presence CME (Central Macular Edema) or PDR (Proliferative Diabetic Retinopathy)

SECONDARY OUTCOMES:
DR severity level | 5 years
  ETDRS grading
Retinal thickness analysis | 5 years
  Retinal thickness (RT) in central subfield, inner and outer rings, assessed by SD-OCT and using layer-by-layer segmentation
Ellipsoid zone analysis | 5 years
  Degree of integrity of the ellipsoid zone, assessed by SD-OCT
Choroidal thickness analysis | 5 years
  Choroidal thickness assessed by Enhanced Depth Imaging (EDI) SD-OCT
SD- OCT- Angiography analysis | 5 years
  Vessel analysis, assessed by SD-OCT OCT-Angiography
OCT-Leakage analysis | 5 years
  LOR (low optical reflectivity) ratio in central subfield, inner and outer ring for assessment of BRB breakdown, assessed by OCT-Leakage
Retinal thickness quantification | 5 years
  Retinal nerve fiber layer thickness (RNFL) and ganglion cells layer (GCL) + inner plexiform layer thickness (IPL) thickness, assessed by layer-by-layer SD-OCT
mfERG assessement | 5 years
  P1 implicit time and P1 amplitude by ring

CONTACTS AND LOCATIONS:
Locations (1):
- Aibili-Cec, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Martinho AC, Marques IP, Messias AL, Santos T, Madeira MH, Sousa DC, Lobo C, Cunha-Vaz J. Ocular and Systemic Risk Markers for Development of Macular Edema and Proliferative Retinopathy in Type 2 Diabetes: A 5-Year Longitudinal Study. Diabetes Care. 2021 Jan;44(1):e12-e14. doi: 10.2337/dc20-1125. Epub 2020 Nov 6. No abstract available. PMID 33158947
- [Derived] Marques IP, Alves D, Santos T, Mendes L, Santos AR, Lobo C, Durbin M, Cunha-Vaz J. Multimodal Imaging of the Initial Stages of Diabetic Retinopathy: Different Disease Pathways in Different Patients. Diabetes. 2019 Mar;68(3):648-653. doi: 10.2337/db18-1077. Epub 2018 Dec 6. PMID 30523027